CLINICAL TRIAL: NCT07013539
Title: Clinical Evaluation of the Efficacy of a Food Supplement in Relieving Premenstrual Syndrome (PMS) Symptoms: a Randomized, Double-blind, Parallel-group, Placebo-controlled Study
Brief Title: Efficacy of a Food Supplement in Relieving Premenstrual Syndrome Symptoms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Activ'inside (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IT00011934/25 Versione n°03
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Premenstrual Syndrome-PMS
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Plant Extracts

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active product (Active Comparator): Hard shell capsule containing active compound.
  Interventions: Dietary Supplement: plant extract
- Control product (Placebo Comparator): Hard shell capsule containing maltodextrine
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: plant extract — hard shell capsule containing plant extract
  Arms: Active product
Dietary Supplement: Placebo — hard shell capsule containing maltodextrine
  Arms: Control product

SUMMARY:
The aim of this clinical trial, funded by Activ'Inside, is to evaluate the efficacy of a food supplement in relieving Premenstrual Syndrome (PMS) Symptoms. The study will be performed on 110 healthy women who experience mild/moderate Premenstrual Syndrome (PMS) symptoms, under the supervision of a board-certified Gynecologist. Half of the subjects will assume the active product and half of the subjects will assume a placebo (a product without active ingredients). Specific assessments will be carried out before and after 1, 2 and 3 menstrual cycles of product intake. Also, the possible occurrence of adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects
* Caucasian ethnicity
* Subjects of childbearing age, between 18 and 45 years (extremes included)
* Subjects who experience mild/moderate Premenstrual Syndrome (PMS) symptoms for at least 3 menstrual cycles prior the beginning of the experimental phase of the study*
* Subjects who have regular menstrual cycles: 21- to 35-day intervals between two menstrual cycles and a menstrual flow duration of 2-8 days**
* Normal weight (BMI greater than or equal to 18.5 to 24.9 kg/m2) ***
* Subjects registered with National Health Service (NHS)
* Subjects certifying the truthfulness of the personal data disclosed to the investigator
* Subjects able to understand the language used in the investigation centre and the information given by the investigator
* Subjects able to respect the instructions given by the investigator as well as able to respect the study constraints and specific requirements
* Commitment not to change the daily routine or the lifestyle
* Stable pharmacological therapy (except for the pharmacological therapy in the non-inclusion criteria) for at least one month without any changes expected or planned during the study
* Subjects informed about the test procedures who have signed a consent form.

  * Assessed by the psychologist using the Premenstrual Symptoms Screening Tool (PSST), a validated self-assessment questionnaire designed to identify women experiencing Premenstrual Syndrome (PMS). The PSST includes questions addressing physical, psychological, and behavioural symptoms. Participants will complete the questionnaire for three consecutive months, and the psychologist will confirm whether they suffer from mild to moderate PMS.

    * Verified by a diary in which participants record this information. Subjects complete the diary for three consecutive months.

      * According to the World Health Organization (WHO) BMI Classification.

Exclusion Criteria:

* Subjects who do not meet the inclusion criteria
* Subjects in the perimenopausal period
* Subjects with any acute, chronic, or progressive disease or condition that may interfere with the study data or that the investigator considers dangerous to the subject or incompatible with the requirements of the study****
* Subjects participating or planning to participate in other clinical trials
* Subjects who participated in a similar study without respecting an adequate washout period (at least one month)
* Subjects that have food intolerances or food allergies to ingredients of the study product
* Subjects under pharmacological treatments that are considered incompatible with the study requirement by the investigator*****
* Subjects who are currently using food supplement(s) and/or products with the same activity as the study product, or who haven't observed an adequate washout period (at least one month)
* Subjects admitted to a health or social facility
* Subjects planning a hospitalization during the study
* Subjects not able to be contacted in case of emergency
* Subjects deprived of freedom by administrative or legal decision or under guardianship
* Subjects with a history of drug, alcohol and other substance abuse
* Subjects with eating disorders (i.e. bulimia, psychogenic eating disorders, etc.)
* Subject breastfeeding, pregnant or not willing to take necessary precautions to avoid pregnancy during the study (for the women of childbearing potential).

  * Polycystic ovary syndrome, endometriosis, thyroid disease, chronic fatigue syndrome, irritable bowel syndrome (IBS), psychiatric disorder (including depression, anxiety, bipolar).

    * Anti-depressants, anxiolytics, diuretics, hormonal contraceptives, nonsteroidal anti-inflammatory drugs.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
PAF-SF | From enrollment to 4, 8, 12 weeks after supplementation
  The Premenstrual Assessment Form Short Form (PAF-SF) is a standardized questionnaire designed to evaluate the severity and impact of premenstrual syndrome (PMS) symptoms. The total score can range from 10 to 60 points, with higher scores indicating greater severity of symptoms.

SECONDARY OUTCOMES:
PHQ-4 | From enrollment to 4, 8, 12 weeks after supplementation
  The Patient Health Questionnaire-4 (PHQ-4) is a brief, validated tool for assessing depression and anxiety symptoms. It consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2). Each item asks how often the individual has been bothered by specific issues over 2 weeks, with responses rated on a scale from 0 (not at all) to 3 (nearly every day). .

OTHER OUTCOMES:
Self-evaluation questionnaire | From enrollment to the end of the treatment at 12 weeks
  The self-evaluation questionnaire consists of 11 questions, and it allows to evaluate the perceived efficacy and pleasantness of the product. The questionnaire consists of multiple-response questions.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rita Mocciaro Specialist in Gynaecology, Principal Investigator
Locations (6):
- Italy (6):
  - Nutratech S.r.l. - Via Francesco Todaro 20/22, Rende, Cosenza
  - Complife Italia S.r.l. - Via Mortara 171, Ferrara, Ferrare
  - Complife Italia S.r.l. - Via Signorelli 159,, Garbagnate Milanese, Milan
  - Complife Italia S.r.l. - Piazzale Siena 11, Milan, Milan
  - Complife Italia SRL - Corso San Maurizio 25, Biella, Pavia
  - Complife Italia SRL- Via Monsignor Angelini 21, San Martino Siccomario, Pavia

IPD SHARING:
Plan to Share IPD: No
confidential data